CLINICAL TRIAL: NCT04902274
Title: Effectiveness of Transcranial Direct Current Stimulation (tDCS) in Musculoskeletal Rehabilitation.
Brief Title: Effectiveness of Transcranial Direct Current Stimulation (tDCS).
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Fellowship Graduation December 2021
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19KACH005
Record Dates: First submitted 2021-05-18; First posted 2021-05-26 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2021-05

CONDITIONS: Ankle Sprains; Musculoskeletal Injury
MeSH Terms: conditions — Ankle Injuries | interventions — Transcranial Direct Current Stimulation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Direct Current Stimulation plus Physical Therapy (Experimental): Participants in the experimental group will receive the current standard of care in ankle inversion sprain rehabilitation plus a 20-minute application of tDCS during each treatment session via the Halo Sport (Halo Neuroscience, San Francisco, CA) headset. The rehabilitation program will be standardized among all patients and will consist of therapeutic exercises, manual physical therapy, and other modalities. Rehabilitation sessions will be performed 2x weekly and sessions will last approximately 45 to 60 minutes.
  Interventions: Other: Transcranial Direct Current Stimulation; Other: Physical Therapy
- Sham Transcranial Direct Current Stimulation plus Physical Therapy (Sham Comparator): Participants in the sham control group will receive the current standard of care in ankle inversion sprain rehabilitation plus a 20-minute sham tDCS treatment, where the patient is wearing the tDCS headset, but stimulation is only applied for 30 seconds of the 20-minute period. The rehabilitation program will be standardized among all patients and will consist of therapeutic exercises, manual physical therapy, and other modalities. Rehabilitation sessions will be performed 2x weekly and sessions will last approximately 45 to 60 minutes.
  Interventions: Other: Sham Transcranial Direct Current Stimulation; Other: Physical Therapy

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation — The Halo Sport (Halo Neuroscience, San Francisco, CA) is a commercial off-the-shelf tDCS device that delivers a 2.2 mA current to the motor cortex through three elastomer foam scalp pads with a 24 sq. cm surface area (see https://www.haloneuro.com/). The tDCS is controlled through the Halo Sport App where the therapist and patient are blind to an actual or sham treatment. Patients in the tDCS group will complete a 20-minute tDCS session while performing the warm-up.
  Arms: Transcranial Direct Current Stimulation plus Physical Therapy
Other: Sham Transcranial Direct Current Stimulation — The Halo Sport (Halo Neuroscience, San Francisco, CA) is a commercial off-the-shelf tDCS device that delivers a 2.2 mA current to the motor cortex through three elastomer foam scalp pads with a 24 sq. cm surface area (see https://www.haloneuro.com/). The tDCS is controlled through the Halo Sport App where the therapist and patient are blind to an actual or sham treatment. Patients in the sham tDCS group will complete a 20-minute sham-tDCS session while performing the warm-up, but the app will discontinue the treatment after 30 seconds.
  Arms: Sham Transcranial Direct Current Stimulation plus Physical Therapy
Other: Physical Therapy — After the tDCS session is complete, the patient will complete treatment consistent with the standard of care for rehabilitation of acute ankle inversion sprain. The rehabilitation program will be standardized among all patients and will consist of therapeutic exercises, manual physical therapy, and other modalities. Rehabilitation sessions will be performed 2x weekly and sessions will last approximately 45 to 60 minutes. Patients will also perform a standardized home exercise program that reinforces the in-clinic treatment.

SUMMARY:
Reducing pain and recovery of strength and function are major challenges in physical therapy. Transcranial direct current stimulation (tDCS) is a novel intervention that has gained popularity in the rehabilitation of athletic injuries, pain management, and sports performance. Acute application of tDCS has been shown to modulate the perception of effort and fatigue, enhance motor learning, improve endurance performance, and improve muscular power and strength. tDCS has also been shown to reduce pain in patients with chronic pain conditions. Using a double-blind, randomized clinical trial design, we aim to evaluate the effectiveness of tDCS plus standard rehabilitation compared to rehabilitation alone on pain, balance and proprioception, functional performance, and strength following acute ankle inversion sprain. We hypothesize that the group using tDCS will demonstrate superior outcomes in all variables of interest.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40
2. Within 2-weeks s/p acute grade 1 or 2 ankle inversion sprain

Exclusion Criteria:

1. Self-Reported Pregnancy
2. Being treated for and on medication for a mental health diagnosis
3. Concussion or non-lateral ankle sprain lower extremity injuries within the past 6 months
4. Open wound or dermatologic lesion on the head or region of application
5. Active implantable medical devices such as cochlear implants or cardiac pacemakers, or with metal implants in the head (excluding standard orthodontic braces, fillings, etc.).
6. Epilepsy or history of seizures
7. Participants who are not fluent in English

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Composite Pain Rating | Change from Baseline to 4-weeks
  Numerical Pain Rating Scale assessment of Current, Best 24-hour, Worst 24-hour Pain
Composite Pain Rating | Change from Baseline to 8-weeks
  Numerical Pain Rating Scale assessment of Current, Best 24-hour, Worst 24-hour Pain

SECONDARY OUTCOMES:
Self-Reported Function | Change from Baseline to 4-weeks
  Patient report of function assessed by Single Assessment Numeric Evaluation
Self-Reported Function | Change from Baseline to 8-weeks
  Patient report of function assessed by Single Assessment Numeric Evaluation
Muscle Strength | Change from Baseline to 4-weeks
  Isometric dorsiflexion, plantarflexion, inversion, eversion assessed by hand-held dynamometry
Muscle Strength | Change from Baseline to 8-weeks
  Isometric dorsiflexion, plantarflexion, inversion, eversion assessed by hand-held dynamometry
Proprioception | Change from Baseline to 4-weeks
  Limits of stability test and unilateral stance test assessed by NeuroCom EquiTest
Proprioception | Change from Baseline to 8-weeks
  Limits of stability test and unilateral stance test assessed by NeuroCom EquiTest
Dynamic balance | Change from Baseline to 4-weeks
  Dynamic balance assessed by the Y-balance Test
Dynamic balance | Change from Baseline to 8-weeks
  Dynamic balance assessed by the Y-balance Test
Muscle Power | Change from Baseline to 4-weeks
  Single leg hop test for distance
Muscle Power | Change from Baseline to 8-weeks
  Single leg hop test for distance

CONTACTS AND LOCATIONS:
Locations (1):
- Keller Army Community Hospital - Arvin Physical Therapy, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No